CLINICAL TRIAL: NCT02912988
Title: A Randomized Trial of Letrozole as an Adjunct to Follicle Stimulating Hormone in Stimulated in Vitro Fertilization Cycles
Brief Title: Letrozole in Stimulated IVF Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 16-014
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2022-11

CONDITIONS: Subfertility
Keywords: Subfertility; In-vitro fertilization; Letrozole
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole group (Experimental): Letrozole + standard treatment:
  Daily 150-300 IU human menopausal gonadotrophin (HMG) / Follicle stimulating hormone (FSH) from cycle day 2-4 (at least 5 days after stopping the oral contraceptive pill) and co-treatment with letrozole 2.5 mg daily from stimulation day 5 until the day before hCG administration. GnRH antagonist (cetrotide or orgalutran) 0.25 mg daily from stimulation day 5 until the day of hCG administration.
  Interventions: Drug: Letrozole
- Control group (No Intervention): Standard treatment:
  Daily 150-300 IU HMG/FSH cycle day 2-4 (at least 5 days after stopping the oral contraceptive pill) until the day before hCG administration. GnRH antagonist 0.25 mg daily from stimulation day 5 until the day of hCG administration.

INTERVENTIONS:
Drug: Letrozole — Daily 150-300 IU human menopausal gonadotrophin (HMG) / Follicle stimulating hormone (FSH) from cycle day 2-4 (at least 5 days after stopping the oral contraceptive pill) and co-treatment with letrozole 2.5 mg daily from stimulation day 5 until the day before hCG administration. GnRH antagonist (cetrotide or orgalutran) 0.25 mg daily from stimulation day 5 until the day of hCG administration.
  Other Names: Letrozole-Teva
  Arms: Letrozole group

SUMMARY:
In-vitro fertilization (IVF) is the treatment of choice for couples with prolonged infertility. The treatment usually involves hormonal stimulation of the ovaries by follicle stimulating hormone (FSH), followed by surgical removal of eggs which are then mixed with sperm in the laboratory to create embryos. The success rates of IVF treatment remain unsatisfactory and are no longer increasing. One of the reasons is an adverse effect of high serum estradiol levels following FSH stimulation on the lining of the uterus.

Letrozole is a drug used in the prevention of recurrence of breast cancer because of its action to reduce the intra-ovarian aromatization of androgens to estrogens. It is now increasingly used for ovulation induction and is as safe as clomiphene citrate. Use of letrozole during standard ovarian stimulation for IVF producing adequate numbers of oocytes with physiological levels of estradiol may increase the present success rate of standard IVF treatment.

The aim of this randomized study is to compare the live birth rate of FSH alone versus combined FSH and letrozole used for ovarian stimulation in IVF treatment.

DETAILED DESCRIPTION:
Trial design:

Infertile women undergoing IVF treatment will be randomized into one of the following two groups by an online randomization program:

Letrozole group: letrozole 2.5mg daily will be given at the start of the antagonist during ovarian stimulation i.e. day 5 of stimulation.

Control group: standard care with FSH alone during ovarian stimulation.

Intervention:

Subjects can be put on oral contraceptive pill in the preceding cycle for scheduling stimulation. On day 2-3, a pelvic ultrasound will be performed for antral follicle count.

Letrozole group:

Daily 150-225 IU human menopausal gonadotrophin (HMG) / Follicle stimulating hormone (FSH) from cycle day 2-4 (at least 5 days after stopping the oral contraceptive pill) and co-treatment with letrozole 2.5 mg daily from stimulation day 5 until the day before hCG administration. GnRH antagonist (cetrotide or orgalutran) 0.25 mg daily from stimulation day 5 until the day of hCG administration.

Control group:

Daily 150-225 IU HMG/FSH cycle day 2-4 (at least 5 days after stopping the oral contraceptive pill) until the day before hCG administration. GnRH antagonist 0.25 mg daily from stimulation day 5 until the day of hCG administration.

A blood sample will be taken and analyzed in the local laboratory for serum E2, P and testosterone levels on cycle day 2 or 3 (baseline) and day of hCG (or the day before). The remaining serum will be frozen and stored for later analysis.

A sample of follicular fluid (FF) will be collected from the first blood free follicle. The FF will be frozen and stored for later analysis: Estradiol, testosterone, inhibin B and AMH levels.

All techniques of IVF including harvesting of oocytes, insemination with specially prepared sperm, embryo culture in the laboratory, embryo transfer and luteal phase support will be according to local protocols. One or two embryos or blastocysts will be replaced.

A pregnancy test will be carried out 2 weeks after embryo transfer in both arms. All women who have a positive pregnancy test 2 weeks after embryo transfer will undergo a transvaginal ultrasound scan to identify the presence and number of gestation sac with a fetal heart signifying an ongoing pregnancy. Pelvic scan will be repeated at 8 weeks, 12 weeks, 24 weeks and 36 weeks of gestation for fetal growth.

ELIGIBILITY:
Inclusion Criteria:

* women under 42 years of age
* medical indication for IVF treatment
* antral follicle count prior to ovarian stimulation >=3
* informed consent

Exclusion Criteria:

* women using donor oocytes
* women undergoing preimplantation genetic diagnosis
* women with abnormal uterine cavity shown on hysterosalpingogram or saline infusion sonogram
* women with hydrosalpinges shown on scanning and not corrected
* previous documented poor response (<=3 oocytes) to ovarian stimulation using at least FSH 225 IU daily

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Live birth rate | through study completion, an average of 1 year
  A baby born alive after 20 weeks gestation

SECONDARY OUTCOMES:
Miscarriage rate | up to 20 weeks of gestation
  Miscarriage before 20 weeks gestation
Clinical and ongoing pregnancy rates | up to 20 weeks
  Presence of at least one gestational sac on ultrasound at 6 weeks and 8-10 weeks
Ovarian hyperstimulation rate | about 1 month
  Ovarian hyperstimulation rate classified according to Royal College of Obstetrics and Gynaecology of the United Kingdom
Total IU of FSH used per cycle | about 2 weeks
  Total IU of FSH used per cycle
Number of follicles > 12 mm on day of hCG (or the day before) | about 2 weeks
  Transvaginal ultrasound performed to measure and the follicles on day of hcG or the day before.
Number of oocytes obtained | On the operation day of transvaginal ultrasound guided oocyte retrieval
  Number of oocyte obtained during the operation of transvaginal ultrasound guided oocyte retrieval
Proportion of oocytes resulting in top quality day 2 (or day 3) embryos according to validated morphological criteria. | 2-3 days after the transvaginal ultrasound guided oocyte retrieval operation
  Proportion of oocytes resulting in top quality day 2 (or day 3) embryos according to validated morphological criteria.
Oocyte fertilization rate | 2-3 days after the transvaginal ultrasound guided oocyte retrieval operation
  Oocyte fertilization rate
Number and quality of embryos obtained | 2-3 days after the transvaginal ultrasound guided oocyte retrieval operation
  Number and quality of embryos obtained
Endometrial thickness on day of hCG (or the day before) | on day of hCG (or the day before)
  Endometrial thickness on day of hCG (or the day before) measured by transvaginal ultrasound
Serum E2 level on day of hCG administration (or the day before) | on day of hCG administration (or the day before)
  Hormonal profile on day of hCG administration (or the day before): serum E2 level
Serum P levels on day of hCG administration (or the day before) | on day of hCG administration (or the day before)
  Hormonal profile on day of hCG administration (or the day before): sSerum P level
Serum testosterone levels on day of hCG administration (or the day before) | on day of hCG administration (or the day before)
  Hormonal profile on day of hCG administration (or the day before):serum testosterone level
Follicular fluid E2 level | On the operation day of transvaginal ultrasound guided oocyte retrieval
  Follicular fluid hormonal profile: E2 level
Follicular fluid testosterone level | On the operation day of transvaginal ultrasound guided oocyte retrieval
  Follicular fluid hormonal profile: testosterone level
Follicular fluid inhibin B level | On the operation day of transvaginal ultrasound guided oocyte retrieval
  Follicular fluid hormonal profile: inhibin B level
Follicular fluid AMH level | On the operation day of transvaginal ultrasound guided oocyte retrieval
  Follicular fluid AMH level
Reported side effects | through study completion, an average of 1 year
Complications of pregnancy | through study completion, an average of 1 year
  small for gestational age, low birth weight, preterm delivery, pre-eclampsia, antepartum haemorrhage, congenital anomaly, perinatal mortality, multiple pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — Department of Obstetrics and Gynaecology, The University of Hong Kong
Locations (2):
- China (2):
  - Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo W, Li HWR, Yang Z, Zeng L, Yang R, Qiao J, Li R, Ng EHY. Live birth after letrozole as an adjunct to follicle-stimulating hormone versus follicle-stimulating hormone alone for ovarian stimulation in in vitro fertilisation cycles-study protocol for a randomised controlled trial. Trials. 2022 Apr 1;23(1):247. doi: 10.1186/s13063-022-06185-0. PMID 35365197